CLINICAL TRIAL: NCT03747588
Title: The Effect and Safety of Comparision Between Minimally-invasive and Open Pancreaticoduodenectomy for Pancreatic Cancer : A Randomized Prospective Trial
Brief Title: The Comparision of Minimally-invasive and Open Pancreaticoduodenectomy for Pancreatic Cancer
Acronym: MIOPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pumch06342
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Carcinoma; Surgery
Keywords: minimally-invasive pancreaticoduodenectomy; open pancreaticoduodenectomy; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally-invasive Pancreaticoduodenectomy (Experimental): MIPD
  Interventions: Procedure: Minimally-invasive pancreaticoduodenectomy
- Open Pancreaticoduodenectomy (Placebo Comparator): OPD
  Interventions: Other: Open pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Minimally-invasive pancreaticoduodenectomy — Minimally-invasive pancreaticoduodenectomy for resection of pancreatic tumor
  Arms: Minimally-invasive Pancreaticoduodenectomy
Other: Open pancreaticoduodenectomy — Open pancreaticoduodenectomy for resection of pancreatic tumor
  Arms: Open Pancreaticoduodenectomy

SUMMARY:
Minimally invasive pancreaticoduodenectomy remains one of the most challenging abdominal procedures. Safety and feasibility remain controversial when comparing minimally-invasive with open pancreaticoduodenectomy, especially for malignant tumors.The aim of this study was to compare minimally invasive and open pancreatoduodenectomy for short-term outcomes and long-term follow-up in a randomized trial.

DETAILED DESCRIPTION:
This study is to compare the efficiency and safety between minimally invasive (including laparoscopic and robotic) and open pancreaticoduodenectomy for pancreatic cancer. We design a prospective randomized study. Patients with malignant pancreatic tumor who underwent pancreatoduodenectomy are recruited to the study. After obtaining informed consent, eligible patients are randomly allocated to minimally-invasive or open group before the operation day. The outcomes evaluated were hospital stay, and blood loss, radicality of surgery, duration of operation and complication rate as well as disease free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18yr, <75yr
* Patients with pancreatic cancer or non-pancreatic cancers (biliary duct cancer or ampullary cancer) who underwent pancreatoduodenectomy
* Preoperative imaging assessment is resectable or borderline resectable

Exclusion Criteria:

* Benign tumors of the head of pancreas
* Enhanced CT diagnosis revealed that the excess of SMV was more than 180 degrees, or distant metastasis.
* conversion to laparotomy because of intraoperative difficulty

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall complications | Up to postoperative 30 days
  The proportion of all complications after operation accounted for the total number of patients
Pancreatic fistula | Up to postoperative 30 days
  The international study group (ISGPF) definition: A drain output of any measurable volume of fluid on or after postoperative day 3 with an amylase content greater than 3 times the serum amylase activity. Three different grades of postoperative fistula (grades A, B, C) are defined according to the clinical impact on the patient's hospital course.
Intra-abdominal bleeding | Up to postoperative 30 days
  The International Study Group of Pancreatic Surgery (ISGPS) definition: Blood loss through abdominal drains or nasogastric tube;hematemesis or melena; clinical deterioration of the patient; unexplained hypotension or tachycardia; or laboratory findings such as a decreasing hemoglobin concentration.
Intra-abdominal infection | Up to postoperative 30 days
  Positive cultures of collection of fluid or blood,or persistent fever necessitating treatment with antibiotics and positive detection in image test.

SECONDARY OUTCOMES:
Length of hospital stay (day) | Up to postoperative 2 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

OTHER OUTCOMES:
progression-free survival | Up to postoperative 5 years
  The period between the beginning of treatment and the observation of disease progression or the occurrence of death for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China